CLINICAL TRIAL: NCT03467529
Title: Evaluation of Full-field Coherence Tomography for ex Vivo Staging and Assessment of Superficial Esophageal Squamous Carcinoma: a Pilot Study
Acronym: OESOCiTy
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0456
Record Dates: First submitted 2017-12-04; First posted 2018-03-16 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Esophagus Cancer
Keywords: Superficial esophageal cancer; Squamous cell cancer; Mini invasive imaging; Pre therapeutic assessment; Optical coherence tomography
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non interventional study — Non interventional study

SUMMARY:
New tools are needed to 1) diagnose and 2) stage early esophageal squamous cell carcinoma (SCC) in order to improve outcomes of this frequent and lethal cancer.

Optical coherence tomography (OCT) is an optical technique, which can image human tissue ex vivo and in vivo with a resolution around 30µm and with a depth of 1mm. Full-field optical coherence tomography (FFOCT) is a new modality, which allows to image an ex vivo specimen with a cellular resolution and to perform 3D reconstruction. This device has never been tested on esophageal specimens.

Therefore, the aim of this non-interventional research is 1) to determine FFOCT diagnostic criteria for SCC and 2) to figure if FFOCT allows the staging of the depth of invasion in SCC.

To achieve these goals, we will image ex vivo 10 specimens of endoscopic resection of SCC (endoscopic mucosal resection (EMR) and submucosal dissection (ESD)) using an FFOCT device and we will compare the results with histological analysis of these specimens.

DETAILED DESCRIPTION:
General study methodology

The study presents the following characteristics:

* Observational
* Non interventional imaging study
* Single-centre
* Not controlled
* Prospective Tests and analysis CRF
* Filled by the investigator
* Data from the medical file of the patient Imaging
* As standard of care
* Before endoscopic resection the lesion will be characterized and pictures will be made using white light endoscopy, magnification techniques and electronic chromoendoscopy
* Immediately after endoscopic resection, the specimen will be prepared, oriented and scanned using the FFOCT device (CE marking)
* Imaging movies will be then reviewed by trained readers and compared to movies of healthy patients, findings will be described
* Imaging movies will be compared to pathology slides

Pathology

* After scanning the specimen will be sent to pathology for analysis
* The pathology slides will be scanned to be kept in the study record together with their interpretation

Study schedule

* Total length of study: 24 months
* Methodology and regulatory: 6 months
* Recruitment period: 1 year
* Recruitment among the patients scheduled for the endoscopic procedure in the operative room
* One single visit = inclusion the day of the procedure
* No follow-up required
* Analyses: 3 months
* Paper writing: 3 months

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and more
* Confirmed diagnosis of SCC based on previous biopsy
* Indication for endoscopic resection
* Patient who has read the information notice and confirmed its willing to participate

Exclusion Criteria:

* Pregnancy
* Any contraindication for endoscopic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients will be recruited by the Clinical investigation center by reviewing the scheduled SCC resections each week. All patients scheduled for an endoscopic resection of SCC will be considered for inclusion in the study. The study itself will take place in the department of gastroenterology. Recruitment within one year of inclusion will be possible because our unit is a regional reference center for interventional endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Concordance between FFOCT findings and pathology based on the Paris classification of superficial esophageal cancer in pathology | Immediately after endoscopic resection (Day 0)
  The principal objective of this study will be reached if:
  * the tumoral lesion is correctly identified in the specimen in FFOCT images
  * and/or the normal esophageal mucosa and submucosal and/or normal vessels are correctly identified in the specimen in FFOCT images
  * in at least 8 specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Coron, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No